CLINICAL TRIAL: NCT01510691
Title: The Influence of Retinal Oxygenation on the Clinical Outcomes in Eyes With Different Vitreoretinal Pathologies After a Successful Vitrectomy
Brief Title: Vitrectomy Retinal Oxygenation
Status: Withdrawn | Type: Observational
Why Stopped: Difficulties in recruiting participants
Sponsor: Stefan Sacu (Other)
Responsible Party: Sponsor-Investigator, Stefan Sacu, Ass Prof Priv Doz Dr, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: VE-Oxygen-28062010
Record Dates: First submitted 2012-01-11; First posted 2012-01-16 (Estimated); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Macular Edema
Keywords: Oxygenation of the retinal vessels; vitroretinal surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Epiretinal membrane
- diabetic macular edema
- vein occlusion

SUMMARY:
Vitrectomy is the common treatment for patients with macular edema secondary to epiretinal membrane. Recently, in eyes with diabetic macular edema or persistent macular edema following retinal vein occlusion, vitrectomy will be increasingly performed as an additional treatment modality. In eyes with impaired oxygen situation vitrectomy may improve the retinal oxygen saturation. However, little information is available about the oxygenation and the blood flow of the retinal vessels after vitroretinal surgery.

Hypoxia is a the major trigger of vascular endothelial growth factor (VEGF), which is in turn the most important factor for the development of macular edema. It is a major issue to improve the oxygen situation and the blood flow of the retina and there are just a few not satisfactory procedures available to overcome this problem. However, vitrectomy would be an adequate therapy for many of these diseases, and it would be an appreciated side effect of the treatment in almost every case.

To investigate the influence of oxygenation and blood flow of the retina on clinical outcomes after a successfully 23 gauge vitrectomy in eyes with epiretinal membrane, persistent macular edema following diabetic retinopathy or retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* male or female, at least 18 years of age.
* ophthalmoscopic evidence of epiretinal membrane scheduled for vitrectomy and membrane peeling.
* persistent diabetic macular edema
* written informed consent
* female patients of childbearing potential must have a negative urine pregnancy test.

Exclusion Criteria:

* uncontrolled systemic disease
* symptoms of a clinically relevant illness in the 3 weeks before the first study day
* any ocular condition that in the opinion of the investigator would be a contraindication for the surgical procedure
* history of glaucoma, aphakie or presence of anterior chamber intraocular lens, choroidal neovascularisation, significant cataract, any ocular infection, - history of pars plana vitrectomy.
* contraindication to pupil dilation.
* need for silicon oil or gas after the surgery
* advanced diabetic retinopathy with vitreoretinal tear and/or bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: 20 patients with macular edema following epiretinal membrane Group 2: 20 patients with persistent diabetic macular edema. Group 3: 20 patients with persistent macular edema following retinal vein occlusion
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinical Data | 6 months
  Visus, OCT
Blood Flow Data | 6 months
  Oxygenation of retinal blood vessles and retinal blood flow

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Opthalmology/Clinical Pharmacology, Vienna, Austria